CLINICAL TRIAL: NCT06413212
Title: Exploratory Study of Precise Therapy for Advanced Tumor Patients With Malignant Hydrothorax or Ascites by Using PTC Drug Sensitivity Testing
Status: Recruiting | Type: Observational
Sponsor: Liu Huang (Other)
Collaborators: Beijing GeneX MedLab Co., Ltd (Industry)
Responsible Party: Sponsor-Investigator, Liu Huang, Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJ-IRB20230704
Record Dates: First submitted 2024-01-14; First posted 2024-05-14 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Lung Cancer; Breast Cancer; Gastric Cancer; Colorectal Cancer
Keywords: PTC: Patient-derived tumor-like cell clusters
MeSH Terms: conditions — Lung Neoplasms; Breast Neoplasms; Stomach Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Malignant effusion
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Case group: Participants who were diagnosed as advanced malignancy and would receive 2 cycles of personal therapy based on PTC drug screening tests.
  Interventions: Diagnostic Test: Patient-derived tumor-like cell clusters (PTC) drug sensitivity testing.

INTERVENTIONS:
Diagnostic Test: Patient-derived tumor-like cell clusters (PTC) drug sensitivity testing. — Fresh malignant effusion samples were collected from advanced malignancy patients for PTC drug sensitivity testing, then assess the accuracy of this diagnostic test by combination and analysis with final clinical outcome.

SUMMARY:
To explore the consistency between result of PTC drug screening tests and actual clinical outcome for patients with advanced malignancy.

DETAILED DESCRIPTION:
This study is anticipated to enroll 55 patients with advanced malignancy, and fresh malignant effusion samples collected from patients would be detected by PTC drug screening. In addition, patients would receive 2 cycles of personal therapy based on results of screening tests. By combining PTC drug sensitivity results with patient's treatment process and clinical feedback, researchers may evaluate the sensitiveness and specificity of PTC drug screening technique in predicting clinical outcome for advanced malignancy patients.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 75 years old, regardless of gender.
2. Score of nutrition risk screening 2002 (NRS2002) is less than 3, NRS20023.
3. Advanced and unresectable malignancy confirmed by biopsy diagnosis.
4. Able to tolerate anti-tumor treatment, and without serious cardiopulmonary and other underlying diseases.
5. Score of eastern cooperative oncology group (ECOG) is not higher than 2, ECOG≤2.
6. Anticipated survival exceed six months.
7. At least one measurable lesions (according to RECIST 1.1)
8. Resistance or intolerance to standard therapy regimens.
9. Signed informed consent form voluntarily.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Have Participated other clinical trials in six months.
3. Severe liver dysfunction.
4. Severe renal dysfunction.
5. Patients with cognitive disorder, mental diseases and terrible compliance.
6. Allergic to known chemotherapeutic agents.
7. Other circumstance not suitable to participate in this trial determined by investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients with malignant effusion, above 18 years of age, at Tongji Hospital, Tongji Medical College of HUST
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2023-08-04 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Complete Response (CR) | up to 12 months
  Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Length is measured in millimeters, refers to RECIST 1.1.
Partial Response (PR) | up to 12 months
  At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Length is measured in millimeters, refers to RECIST.1.1.
Progressive Disease (PD) | up to 12 months
  At least a 20% increase in the sum of diameters of taraet lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm (the appearance of one or more new lesions is also considered progression). Length is measured in millimeters, refers to RECIST 1.1.
Stable Disease (SD) | up to 12 months
  Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. Length is measured in millimeters, refers to RECIST 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Liu Huang, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

REFERENCES:
- [Background] Lim ZF, Ma PC. Emerging insights of tumor heterogeneity and drug resistance mechanisms in lung cancer targeted therapy. J Hematol Oncol. 2019 Dec 9;12(1):134. doi: 10.1186/s13045-019-0818-2. PMID 31815659
- [Background] Leonetti A, Sharma S, Minari R, Perego P, Giovannetti E, Tiseo M. Resistance mechanisms to osimertinib in EGFR-mutated non-small cell lung cancer. Br J Cancer. 2019 Oct;121(9):725-737. doi: 10.1038/s41416-019-0573-8. Epub 2019 Sep 30. PMID 31564718
- [Background] Passaro A, Janne PA, Mok T, Peters S. Overcoming therapy resistance in EGFR-mutant lung cancer. Nat Cancer. 2021 Apr;2(4):377-391. doi: 10.1038/s43018-021-00195-8. Epub 2021 Apr 15. PMID 35122001
- [Background] Doroshow DB, Sanmamed MF, Hastings K, Politi K, Rimm DL, Chen L, Melero I, Schalper KA, Herbst RS. Immunotherapy in Non-Small Cell Lung Cancer: Facts and Hopes. Clin Cancer Res. 2019 Aug 1;25(15):4592-4602. doi: 10.1158/1078-0432.CCR-18-1538. Epub 2019 Mar 1. PMID 30824587
- [Background] Wojas-Krawczyk K, Kalinka E, Grenda A, Krawczyk P, Milanowski J. Beyond PD-L1 Markers for Lung Cancer Immunotherapy. Int J Mol Sci. 2019 Apr 18;20(8):1915. doi: 10.3390/ijms20081915. PMID 31003463
- [Background] Reck M, Remon J, Hellmann MD. First-Line Immunotherapy for Non-Small-Cell Lung Cancer. J Clin Oncol. 2022 Feb 20;40(6):586-597. doi: 10.1200/JCO.21.01497. Epub 2022 Jan 5. PMID 34985920
- [Background] Blackley EF, Loi S. Targeting immune pathways in breast cancer: review of the prognostic utility of TILs in early stage triple negative breast cancer (TNBC). Breast. 2019 Nov;48 Suppl 1:S44-S48. doi: 10.1016/S0960-9776(19)31122-1. PMID 31839159
- [Background] Wang X, Wang SS, Huang H, Cai L, Zhao L, Peng RJ, Lin Y, Tang J, Zeng J, Zhang LH, Ke YL, Wang XM, Liu XM, Chen QJ, Zhang AQ, Xu F, Bi XW, Huang JJ, Li JB, Pang DM, Xue C, Shi YX, He ZY, Lin HX, An X, Xia W, Cao Y, Guo Y, Su YH, Hua X, Wang XY, Hong RX, Jiang KK, Song CG, Huang ZZ, Shi W, Zhong YY, Yuan ZY; South China Breast Cancer Group (SCBCG). Effect of Capecitabine Maintenance Therapy Using Lower Dosage and Higher Frequency vs Observation on Disease-Free Survival Among Patients With Early-Stage Triple-Negative Breast Cancer Who Had Received Standard Treatment: The SYSUCC-001 Randomized Clinical Trial. JAMA. 2021 Jan 5;325(1):50-58. doi: 10.1001/jama.2020.23370. PMID 33300950
- [Background] Yamaguchi K, Yoshida K, Tanahashi T, Takahashi T, Matsuhashi N, Tanaka Y, Tanabe K, Ohdan H. The long-term survival of stage IV gastric cancer patients with conversion therapy. Gastric Cancer. 2018 Mar;21(2):315-323. doi: 10.1007/s10120-017-0738-1. Epub 2017 Jun 14. PMID 28616743
- [Background] Pozzo C, Basso M, Cassano A, Quirino M, Schinzari G, Trigila N, Vellone M, Giuliante F, Nuzzo G, Barone C. Neoadjuvant treatment of unresectable liver disease with irinotecan and 5-fluorouracil plus folinic acid in colorectal cancer patients. Ann Oncol. 2004 Jun;15(6):933-9. doi: 10.1093/annonc/mdh217. PMID 15151951
- [Background] Alberts SR, Horvath WL, Sternfeld WC, Goldberg RM, Mahoney MR, Dakhil SR, Levitt R, Rowland K, Nair S, Sargent DJ, Donohue JH. Oxaliplatin, fluorouracil, and leucovorin for patients with unresectable liver-only metastases from colorectal cancer: a North Central Cancer Treatment Group phase II study. J Clin Oncol. 2005 Dec 20;23(36):9243-9. doi: 10.1200/JCO.2005.07.740. Epub 2005 Oct 17. PMID 16230673
- [Background] Falcone A, Ricci S, Brunetti I, Pfanner E, Allegrini G, Barbara C, Crino L, Benedetti G, Evangelista W, Fanchini L, Cortesi E, Picone V, Vitello S, Chiara S, Granetto C, Porcile G, Fioretto L, Orlandini C, Andreuccetti M, Masi G; Gruppo Oncologico Nord Ovest. Phase III trial of infusional fluorouracil, leucovorin, oxaliplatin, and irinotecan (FOLFOXIRI) compared with infusional fluorouracil, leucovorin, and irinotecan (FOLFIRI) as first-line treatment for metastatic colorectal cancer: the Gruppo Oncologico Nord Ovest. J Clin Oncol. 2007 May 1;25(13):1670-6. doi: 10.1200/JCO.2006.09.0928. PMID 17470860
- [Background] Vlachogiannis G, Hedayat S, Vatsiou A, Jamin Y, Fernandez-Mateos J, Khan K, Lampis A, Eason K, Huntingford I, Burke R, Rata M, Koh DM, Tunariu N, Collins D, Hulkki-Wilson S, Ragulan C, Spiteri I, Moorcraft SY, Chau I, Rao S, Watkins D, Fotiadis N, Bali M, Darvish-Damavandi M, Lote H, Eltahir Z, Smyth EC, Begum R, Clarke PA, Hahne JC, Dowsett M, de Bono J, Workman P, Sadanandam A, Fassan M, Sansom OJ, Eccles S, Starling N, Braconi C, Sottoriva A, Robinson SP, Cunningham D, Valeri N. Patient-derived organoids model treatment response of metastatic gastrointestinal cancers. Science. 2018 Feb 23;359(6378):920-926. doi: 10.1126/science.aao2774. PMID 29472484
- [Background] Yin S, Xi R, Wu A, Wang S, Li Y, Wang C, Tang L, Xia Y, Yang D, Li J, Ye B, Yu Y, Wang J, Zhang H, Ren F, Zhang Y, Shen D, Wang L, Ying X, Li Z, Bu Z, Ji X, Gao X, Jia Y, Jia Z, Li N, Li Z, Ji JF, Xi JJ. Patient-derived tumor-like cell clusters for drug testing in cancer therapy. Sci Transl Med. 2020 Jun 24;12(549):eaaz1723. doi: 10.1126/scitranslmed.aaz1723. PMID 32581131